CLINICAL TRIAL: NCT07097025
Title: Efficacy and Safety of Vagus Nerve Stimulation Treatment in Treatment Resistant Depression
Brief Title: 2-Year Study of Vagus Nerve Stimulation for Higher-Grade Treatment-Resistant Depression: Clinical Outcomes and Policy Recommendation
Acronym: VNS TRD HG-TRD
Status: Completed | Type: Observational
Sponsor: Dr.Yoav Domany (Other)
Collaborators: Lev HaSharon Mental Health Center (Unknown); Maaynei Hayesha Medical Center (Other)
Responsible Party: Sponsor-Investigator, Dr.Yoav Domany, Psychiatrist, Department Manager, Maaynei Hayesha Medical Center
Organization: Maaynei Hayesha Medical Center (Other)
Other Study IDs: 0371-23-SMC
Record Dates: First submitted 2025-07-24; First posted 2025-07-31 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Treatment Resistant Depression (TRD); Depression - Major Depressive Disorder; Bipolar Depression
Keywords: TRD; VNS; MDD; Suicidality; depression; policy
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant; Bipolar Disorder; Suicidal Ideation; Depression | interventions — Vagus Nerve Stimulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Treatment Resistant Depression (TRD) patients: Participants were recruited under the care of the participating physician investigators, from the Advanced Treatments for Treatment Resistant Depression (TRD) Clinics at Sheba Medical Center, or Lev-Hasharon mental health center , who underwent VNS implantation procedure.
  Inclusion criteria were age ≥ 18 years; Diagnose of chronic and recurrent depressive episode lasting at least two years (persistent depressive disorder) or a history of at least three depressive episodes, including the current episode, according to the Diagnostic and Statistical Manual of Mental Disorders, fifth edition (DSM-5) criteria; Resistance to treatment was defined as failure to respond to at least four antidepressant treatments, including pharmacotherapy (administered at therapeutic dosages for at least four weeks), psychotherapy, ECT, or esketamine meaning HD-TRD; Baseline scores >20 according to the Montgomery-Åsberg Depression Rating Scale (MADRS)(indicating moderate (20-34) to severe (>34) depression).
  Interventions: Device: vagus nerve stimulation

INTERVENTIONS:
Device: vagus nerve stimulation — VNS is a neuromodulatory treatment involving implantation of a subcutaneous device that delivers intermittent electrical stimulation to the vagus nerve, modulating central pathways associated with mood regulation.
  Other Names: VNS

SUMMARY:
The goal of this observational study is to evaluate whether vagus nerve stimulation (VNS) intervention can reduce depressive symptoms and suicidality in adults with higher-grade treatment-resistant depression (HG-TRD)-individuals who have not responded to at least four prior depression treatments.

The main questions it aims to answer are: does VNS lead to a meaningful and sustained reduction in depression severity over 24 months? and does VNS reduce suicidal thoughts and behaviors in this population?

Participants in this study were adults (age ≥ 18) with chronic or recurrent depression and at least four failed prior treatments, including medication, psychotherapy, electroconvulsive therapy (ECT), or esketamine. They underwent surgical implantation of a VNS device and their depressive symptoms and suicidality assessed at baseline, and then again at 6, 12, 18, and 24 months using the Montgomery-Åsberg Depression Rating Scale (MADRS). The study includes continous follow-upvisits and VNS device adjustments for 2 years post implantation. with outcomes including treatment response, remission, changes in suicidal ideation, and psychiatric hospitalization days over the study period

DETAILED DESCRIPTION:
This prospective, multi-center observational study aimed to evaluate the long-term real-world effectiveness, safety, and clinical utility of vagus nerve stimulation (VNS) in individuals diagnosed with higher-grade treatment-resistant depression (HG-TRD), defined by failure to respond to at least four adequate therapeutic interventions. The study was conducted in three Israeli psychiatric centers between 2020 and 2025.

Vagus nerve stimulation (VNS) is a neuromodulation therapy involving the surgical implantation of a device that delivers electrical stimulation to the vagus nerve, targeting brain regions associated with mood regulation. While VNS is approved in several countries for treatment-resistant depression (TRD), real-world data outside of structured clinical trials for TRD remain limited. This study sought to fill that gap, particularly in the Israeli healthcare context.

Study Population and Procedures

Eligible participants were adults with chronic or recurrent major depressive episodes, who had previously failed at least four depression treatments (e.g., pharmacotherapy, Electro-Convulsive Treatment (ECT), esketamine, psychotherapy). Participants underwent VNS implantation and were followed prospectively for 24 months. Follow-up assessments were conducted at 6, 12, 18, and 24 months, evaluating depression severity, suicidality, and adverse effects using standardized clinical tool, the Montgomery-Åsberg Depression Rating Scale (MADRS).

Device programming and stimulation adjustments were conducted biweekly in the early phases post-implantation and subsequently as clinically indicated. Stimulation parameters were titrated based on clinical response and tolerability.

Data were collected in dedicated TRD specialty clinics and recorded by trained raters using structured clinical forms. All assessments were performed in-person during scheduled follow-up visits.

The study was approved by the institutional Helsinki committees at all participating sites. Written informed consent was obtained from all participants.

Statistical Plan and Handling of Data:

* Sample Size: The final sample included 16 participants who completed 24-month follow-up and were eligible for efficacy analyses. All 19 implanted patients were included in safety analyses.
* Primary analysis involved repeated measures ANOVA to examine changes in MADRS total scores over time.
* Categorical outcomes (response, remission, partial response) were computed at each time-point and cumulatively (best outcome achieved at any time).
* Suicidality was analyzed via MADRS item 10, both as a continuous and categorical outcome (≥50% or ≥30% reduction).
* Hospitalization burden was analyzed as an exploratory outcome, comparing inpatient days during three time intervals (pre-implantation, year 1 post-implantation, year 2 post-implantation).
* Missing data: Participants who permanently deactivated the device within the first 6 months were excluded from efficacy analyses but retained for safety reporting. Missing values in the MADRS and item 10 of this tool (suicidality) were imputed using the last observation carried forward method. Imputation was performed in the case of a missing value between two measurement points, but was not done after the last measurement point (for example, if a participant had values up to month 12, imputing was not done for month 18).

Safety Assessment:

Adverse events were monitored throughout the study and including voice alteration, throat discomfort, and coughing, as well as rarer complications such as dysphagia or transient vocal cord paresis. All adverse events were documented in accordance with clinical research guidelines.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years.
* Diagnose of chronic and recurrent depressive episode lasting at least two years (persistent depressive disorder) or a history of at least three depressive episodes, including the current episode, according to the Diagnostic and Statistical Manual of Mental Disorders, fifth edition (DSM-5) criteria.
* Resistance to treatment was defined as failure to respond to at least four antidepressant treatments, including pharmacotherapy (administered at therapeutic dosages for at least four weeks), psychotherapy, Electroconvulsive treatment (ECT), or esketamine meaning HD-TRD.
* Baseline scores >20 according to the Montgomery-Åsberg Depression Rating Scale (MADRS) (indicating moderate (20-34) to severe (>34) depression).

Exclusion Criteria:

* Lifetime history of psychotic disorders (e.g., schizophrenia, schizoaffective disorder and other) or psychotic features during the current depressive episode.
* Lifetime history of rapid-cycling bipolar disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants were recruited under the care of the participating physician investigators, from the Advanced Treatments for TRD Clinics at Sheba Medical Center (n=10, 62.5% of participants), or and Lev-Hasharon mental health center (n=6, 37.5% of participants).
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Change in Depression Severity (MADRS Total Score) | Baseline to 24 months post-implantation
  Change in depressive symptom severity, as measured by the Montgomery-Åsberg Depression Rating Scale (MADRS) total score. The scale consists of 10 clinician-rated items, each scored from 0 to 6, with total scores ranging from 0 (no symptoms) to 60 (severe depression). A reduction in score indicates clinical improvement. Depression severity was assessed at baseline and at predefined follow-up visits (6, 12, 18, and 24 months post-implantation). The primary outcome reflects the magnitude and trajectory of change in MADRS scores over time following vagus nerve stimulation (VNS) implantation.

SECONDARY OUTCOMES:
Change in Suicidality (MADRS Item 10 Score) | Baseline to 24 months post-implantation
  Change in suicidality as measured by item 10 of the Montgomery-Åsberg Depression Rating Scale (MADRS), which assesses suicidal thoughts and behaviors on a 0-6 scale. A reduction in score indicates clinical improvement. The outcome captures both point-in-time and cumulative reductions in suicidality over the course of 24 months following vagus nerve stimulation (VNS) implantation.
Rates of Remission, Response, and Partial Response | 6 to 24 months post-implantation
  Proportion of participants achieving clinical improvement at predefined follow-up timepoints (6, 12, 18, and 24 months) and cumulatively (i.e., best outcome achieved at any point during follow-up), based on changes in the Montgomery-Åsberg Depression Rating Scale (MADRS) total score:
  * Remission: MADRS total score ≤12
  * Response: ≥50% reduction in MADRS total score from baseline
  * Partial Response: 30%-49% reduction in MADRS total score from baseline
  Each participant was categorized based on the highest level of improvement attained at each timepoint. These outcomes reflect clinically meaningful levels of symptom reduction following vagus nerve stimulation (VNS) implantation.
Safety - Incidence and Nature of Adverse Events | Baseline to 24 months post-implantation
  Incidence, type, severity, and time course of adverse events related to VNS implantation and stimulation, including surgical complications and stimulation-related side effects. Adverse events were documented throughout the 24-month follow-up period and categorized by clinical severity (e.g., mild, moderate, serious), duration, and management strategies (e.g., stimulation adjustment, discontinuation).

OTHER OUTCOMES:
Change in Psychiatric Hospitalization Days | 1 year pre-implantation to 2 years post-implantation
  Change in the number of psychiatric inpatient hospitalization days before and after VNS implantation. Hospitalization burden was calculated for each participant across three time intervals: (1) 12 months pre-implantation, (2) first 12 months post-implantation, and (3) second 12 months post-implantation. Mean hospitalization days per period were compared to assess potential reductions in inpatient care burden following VNS therapy.

CONTACTS AND LOCATIONS:
Locations (2):
- Israel (2):
  - Maaynei Hayeshua medical center, Bnei Brak
  - Lev Hasharon Medical Center, Netanya

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data (IPD) might not be shared due to concerns regarding participant confidentiality and the sensitive nature of the clinical data. The study involves a small cohort of individuals with severe, treatment-resistant depression, and the risk of re-identification cannot be fully mitigated, even with de-identification procedures.

REFERENCES:
- [Background] Rush AJ, Conway CR, Aaronson ST, George MS, Riva-Posse P, Dunner DL, Zajecka J, Bunker MT, Quevedo J, Allen RM, Alva G, Luing H, Nahas Z, Manu L, Bennett JI, Mickey BJ, Becker J, Sheline Y, Cusin C, Murrough JW, Reeves K, Rosenquist PB, Lee YL, Majewski S, Way J, Olin B, Sackeim HA. Effects of vagus nerve stimulation on daily function and quality of life in markedly treatment-resistant major depression: Findings from a one-year, randomized, sham-controlled trial. Brain Stimul. 2025 May-Jun;18(3):690-700. doi: 10.1016/j.brs.2024.12.1187. Epub 2024 Dec 18. PMID 39701918
- [Background] Aaronson ST, Sears P, Ruvuna F, Bunker M, Conway CR, Dougherty DD, Reimherr FW, Schwartz TL, Zajecka JM. A 5-Year Observational Study of Patients With Treatment-Resistant Depression Treated With Vagus Nerve Stimulation or Treatment as Usual: Comparison of Response, Remission, and Suicidality. Am J Psychiatry. 2017 Jul 1;174(7):640-648. doi: 10.1176/appi.ajp.2017.16010034. Epub 2017 Mar 31. PMID 28359201
- [Background] Rush AJ, Conway CR, Aaronson ST. Cost-effectiveness of VNS therapy for difficult-to-treat depression: insights from the RECOVER trial. J Affect Disord. 2024. In Press.
- [Background] Conway CR, Aaronson ST, Greenberg BD, Carpenter LL, Holbert RC, Bunker M, et al. RECOVER VNS Depression Study: One-year outcomes of a randomized, controlled trial. Biol Psychiatry. 2024. In Press.
- [Background] Lynch F, Law CW, McIntyre RS. Vagus nerve stimulation for treatment-resistant depression: efficacy, side effects, and future prospects. CNS Drugs. 2022;36(10):1041-55.
- [Background] Cusin C, Dougherty DD. Somatic therapies for treatment-resistant depression: ECT, TMS, VNS, DBS. Biol Mood Anxiety Disord. 2012 Aug 17;2:14. doi: 10.1186/2045-5380-2-14. PMID 22901565
- [Background] Strawbridge R, Carter B, Marwood L, Bandelow B, Tsapekos D, Nikolova VL, Taylor R, Mantingh T, de Angel V, Patrick F, Cleare AJ, Young AH. Augmentation therapies for treatment-resistant depression: systematic review and meta-analysis. Br J Psychiatry. 2019 Jan;214(1):42-51. doi: 10.1192/bjp.2018.233. Epub 2018 Nov 20. PMID 30457075
- [Background] Rush AJ, Sackeim HA, Conway CR, Bunker MT, Hollon SD, Demyttenaere K, Young AH, Aaronson ST, Dibue M, Thase ME, McAllister-Williams RH. Clinical research challenges posed by difficult-to-treat depression. Psychol Med. 2022 Feb;52(3):419-432. doi: 10.1017/S0033291721004943. Epub 2022 Jan 7. PMID 34991768
- [Background] Lam RW, Milev R, Rotzinger S, Andreazza AC, Blier P, Brenner C, et al. Canadian Network for Mood and Anxiety Treatments (CANMAT) 2023 Clinical Guidelines for the Management of Adults with Major Depressive Disorder: Section 5. Difficult-to-treat depression. Can J Psychiatry. 2024;69(2):95-120.
- [Background] McAllister-Williams RH, Arango C, Blier P, Demyttenaere K, Falkai P, Gorwood P, Hopwood M, Javed A, Kasper S, Malhi GS, Soares JC, Vieta E, Young AH, Papadopoulos A, Rush AJ. The identification, assessment and management of difficult-to-treat depression: An international consensus statement. J Affect Disord. 2020 Apr 15;267:264-282. doi: 10.1016/j.jad.2020.02.023. Epub 2020 Feb 7. PMID 32217227
- [Background] Perez-Sola V, Roca M, Alonso J, Gabilondo A, Hernando T, Sicras-Mainar A, Sicras-Navarro A, Herrera B, Vieta E. Economic impact of treatment-resistant depression: A retrospective observational study. J Affect Disord. 2021 Dec 1;295:578-586. doi: 10.1016/j.jad.2021.08.036. Epub 2021 Aug 27. PMID 34509073
- [Background] Fava M. Diagnosis and definition of treatment-resistant depression. Biol Psychiatry. 2003 Apr 15;53(8):649-59. doi: 10.1016/s0006-3223(03)00231-2. PMID 12706951
- [Background] Otte C, Gold SM, Penninx BW, Pariante CM, Etkin A, Fava M, Mohr DC, Schatzberg AF. Major depressive disorder. Nat Rev Dis Primers. 2016 Sep 15;2:16065. doi: 10.1038/nrdp.2016.65. PMID 27629598